CLINICAL TRIAL: NCT01322347
Title: A Randomized, Placebo-Controlled, Phase III Study of Dialysate Containing Soluble Ferric Pyrophosphate (SFP) in Chronic Kidney Disease Patients Receiving Hemodialysis: The Continuous Replacement Using Iron Soluble Equivalents (CRUISE 2) Study
Brief Title: Continuous Soluble Ferric Pyrophosphate (SFP) Iron Delivery Via Dialysate in Hemodialysis Patients (CRUISE 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMTI-SFP-5
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: End Stage Renal Disease; Hemodialysis; SFP; Hemodialysis-dependent chronic renal failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soluble Ferric Pyrophosphate (SFP) in dialysate (Active Comparator): 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Interventions: Drug: Soluble Ferric Pyrophosphate (SFP)
- Standard Dialysate (Placebo Comparator): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Interventions: Device: Standard dialysate

INTERVENTIONS:
Drug: Soluble Ferric Pyrophosphate (SFP) — Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 18 months.
  Arms: Soluble Ferric Pyrophosphate (SFP) in dialysate
Device: Standard dialysate — Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week.
  Arms: Standard Dialysate

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Soluble Ferric Pyrophosphate (SFP) dialysate solution in maintaining iron delivery for erythropoiesis in anemic adult patients with chronic kidney disease (CKD) receiving hemodialysis. Efficacy will be measured primarily by the change from baseline in hemoglobin (Hgb).

DETAILED DESCRIPTION:
Screening: 2-3 weeks prior to enrollment in Stage 1.

Stage 1 (Run-In): 1-4weeks depending on qualification for Stage 2.

Stage 2 (Randomized Blinded Treatment): 12 months unless withdrawn prematurely.

Stage 3 (Open-Label Treatment): The duration of Stage 2 plus Stage 3 is intended to be 18 months regardless of treatment assignment in Stage 2.

ELIGIBILITY:
Stage 1:

Main Inclusion Criteria:

* Adult subject ≥ 18 years of age undergoing chronic hemodialysis three or four times per week for chronic kidney disease (CKD) for at least 4 months, and expected to remain on hemodialysis three to four times weekly and be able to complete the duration of the study.
* Received IV iron therapy between 6 months and 2 weeks prior to enrollment in order to replace iron losses resulting from hemodialysis procedure.
* Mean Screening Hgb ≥ 9.5 to ≤ 11.5 grams per deciliter (g/dL).
* Mean Screening Transferrin Saturation (TSAT) ≥ 15% to ≤ 40%.
* Mean Screening serum ferritin ≥ 200 to ≤ 800 micrograms per liter (µg/L).
* If being administered epoetin, darbepoetin, or CERA, epoetin dose ≤ 45,000 Units (U)/week, darbepoetin dose ≤ 200 micrograms (µg)/week, or CERA dose ≤ 400 micrograms (µg)/month during the four weeks prior to enrollment.

Main Exclusion Criteria:

* Patient has living kidney donor identified or living-donor kidney transplant scheduled. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
* Vascular access for dialysis with femoral catheter or non-tunneled catheter.
* Received a total of > 800 milligrams (mg) IV iron during the 8 weeks prior to enrollment.
* If being administered an ESA, route of administration change or ESA dose change > 35% (i.e., [max - min dose]/max dose > 0.35) over the 2 weeks prior to screening.
* Serum albumin < 3.0 grams per deciliter (g/dL) any time over the 8 weeks prior to enrollment.
* Red Blood Cell (RBC) or whole blood transfusion within 12 weeks prior to enrollment.

Stage 2:

Main Inclusion Criteria:

* Patient currently enrolled in the Stage 1 run-in period of study.
* Undergoing chronic hemodialysis three or four times per week for chronic kidney disease (CKD), and expected to remain on hemodialysis three to four times weekly and be able to complete duration of the study.
* Mean Hgb ≥ 9.5 to ≤ 11.5 g/dL over the three most recent consecutive every-week measurements prior to randomization.
* Stable Hgb defined as ≤ 1.0 g/dL difference between the maximum and minimum Hgb values over the 3 weeks immediately prior to randomization.
* Mean TSAT ≥ 15% to ≤ 40% over the two most recent consecutive every-other-week measurements prior to randomization.
* Mean serum ferritin ≥ 200 to ≤ 800 µg/L over the two most recent consecutive every-other-week measurements prior to randomization.
* If being administered epoetin, darbepoetin, or CERA, epoetin dose ≤ 45,000 U/week, darbepoetin dose ≤ 200 µg/week, or CERA dose ≤ 400 µg/month during the four weeks prior to randomization.

Main Exclusion Criteria:

* Patient has living kidney donor identified or living-donor kidney transplant scheduled. (Note: Patients awaiting deceased-donor transplant need not be excluded.)
* Vascular access for dialysis with femoral catheter or non-tunneled catheter.
* Received any amount of IV iron during the 4 weeks prior to randomization.
* If being administered an (Erythropoietin Stimulating Agent) ESA, change in dose over the 6 weeks immediately prior to randomization.
* Serum albumin < 3.0 g/dL any time over the 8 weeks prior to randomization.
* RBC or whole blood transfusion during Stage 1.

Stage 3:

Main Inclusion Criteria:

* Patient randomized in Stage 2 who has completed the full duration of Stage 2 and less than 4 weeks have elapsed since completion of Stage 2, OR
* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for protocol-defined Protocol-Mandated Change in Anemia Management and less than 4 weeks have elapsed since withdrawal from Stage 2, OR
* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for Hgb >11.5 g/dL over ≥ 1 week confirmed by ≥ 2 consecutive measurements AND an associated increase in Hgb by ≥ 1 g/dL over 4 weeks.

Main Exclusion Criteria:

* Patient in Stage 2 who has been prematurely withdrawn from Stage 2 for any reason other than as noted in inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray Pratt, MD, Study Director — Rockwell Medical
Locations (36):
- United States (34):
  - Investigator, Paragould, Arkansas
  - Investigator, Pine Bluff, Arkansas
  - Investigator, Alhambra, California
  - Investigator, Beverly Hills, California
  - Investigator, Glendale, California
  - Investigator, La Mesa, California
  - Investigator, Long Beach, California
  - Investigator, Lynwood, California
  - Investigator, Paramount, California
  - Investigator, Whittier, California
  - Investigator, Pembroke Pines, Florida
  - Investigator, Augusta, Georgia
  - Investigator, Macon, Georgia
  - Investigator, Meridian, Idaho
  - Investigator, Hines, Illinois
  - Investigator, Rockville, Maryland
  - Investigator, Detroit, Michigan
  - Investigator, Pontiac, Michigan
  - Investigator, Southfield, Michigan
  - Investigator, Eatontown, New Jersey
  - Investigator, Brooklyn, New York
  - Investigator, Fresh Meadows, New York
  - Investigator, Great Neck, New York
  - Investigator, Orchard Park, New York
  - Investigator, The Bronx, New York
  - Investigator, Bethany, Oklahoma
  - Investigator, Bethlehem, Pennsylvania
  - Investigator, Philadelphia, Pennsylvania
  - Investigator, Nashville, Tennessee
  - Investigator, Arlington, Texas
  - Investigator, Fort Worth, Texas
  - Investigator, Houston, Texas
  - Investigator, San Antonio, Texas
  - Investigator, Fairfax, Virginia
- Canada (2):
  - Investogator, Edmonton, Alberta
  - Investigator, Greenfield Park, Quebec

REFERENCES:
- [Derived] Fishbane SN, Singh AK, Cournoyer SH, Jindal KK, Fanti P, Guss CD, Lin VH, Pratt RD, Gupta A. Ferric pyrophosphate citrate (Triferic) administration via the dialysate maintains hemoglobin and iron balance in chronic hemodialysis patients. Nephrol Dial Transplant. 2015 Dec;30(12):2019-26. doi: 10.1093/ndt/gfv277. Epub 2015 Jul 13. PMID 26175145

RESULTS

PARTICIPANT FLOW:
Groups:
- Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 48 weeks.
- Standard Dialysate (Placebo): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 48 weeks.
Period: Overall Study
Arm/Group | Soluble Ferric Pyrophosphate (SFP) in Dialysate | Standard Dialysate (Placebo)
Started | 147 | 147
Completed 48 Wks in St 2 | 28 | 22
Comp St 2 Due to ESA/IV Iron Needs | 68 | 90
Enrolled in St 3 | 101 | 113
Completed St 3 | 82 | 86
Completed | 96 | 112
Not Completed | 51 | 35
Not completed — Adverse Event | 7 | 2
Not completed — Death | 5 | 3
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 5 | 2
Not completed — Withdrawal by Subject | 1 | 4
Not completed — non-protocol change to ESA or IV iron | 14 | 6
Not completed — blood transfusion | 5 | 5
Not completed — sponsor decision | 1 | 3
Not completed — ineligible | 6 | 3
Not completed — kidney transplant | 3 | 1
Not completed — study drug withheld > 12 wks | 0 | 1
Not completed — moved/changed dialysis | 2 | 4

BASELINE CHARACTERISTICS:
Population: intent-to-treat: all randomized subjects, regardless of whether they received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Soluble Ferric Pyrophosphate (SFP) in Dialysate | Standard Dialysate (Placebo) | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.68) | 59.0 (14.38) | 58.5 (13.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 54 | 119
  Male | 82 | 93 | 175
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 36 | 69
  Not Hispanic or Latino | 114 | 111 | 225
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 64 | 54 | 118
  White | 73 | 83 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 128 | 123 | 251
  Canada | 19 | 24 | 43
Height [Mean (Standard Deviation); unit: centimeters] | 168.80 (10.238) | 170.01 (9.944) | 169.40 (10.093)
Post-dialysis weight [Mean (Standard Deviation); unit: kilograms] | 86.64 (22.270) | 85.09 (23.474) | 85.86 (22.857)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hemoglobin at End-of-Treatment: Least-Squares Mean
Description: Mean change from baseline Hgb (the average of the three most recent Hgb values preceding randomization) assessments during the last one-sixth of the treatment period for patients who prematurely withdraw from study treatment, but will include a minimum of at least the last two Hgb values. Value is expressed as least-squares mean, along with standard error.
Time Frame: Hgb measured weekly; up to 48 weeks from date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study drug and had at least one post-dose hemoglobin value measured.
Measure: Least Squares Mean (Standard Error); unit: grams per liter
Groups:
- Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week for up to 48 weeks.
- Stage 2 Placebo (Standard Dialysate): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week for up to 48 weeks.
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
grams per liter | -0.5 (1.08) | -4.0 (1.09)
Statistical Analysis 1: Comparison: Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate vs Stage 2 Placebo (Standard Dialysate); Test type: Superiority or Other; p = 0.011, ANCOVA — LS Mean (SE) and p-value are from ANCOVA model with baseline Hgb as covariate. Model also includes indicator variable for baseline ESA dose stratum; Difference in LS Means between SFP & PBO = 3.6, Standard Error of Mean 1.39

2. Secondary Outcome: Mean Change in Serum Iron From Pre-Dialysis to Post-Dialysis
Description: The mean difference between the pre-dialysis and post-dialysis serum iron was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study drug and had at least one post-dialysis hemoglobin measured.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
micromoles per liter
  mean pre-dialysis serum iron | 11.634 (3.2506) | 11.086 (3.0143)
  mean post-dialysis serum iron | 31.347 (7.9885) | 12.247 (4.0720)
  serum iron change from pre- to post-dialysis | 19.675 (6.8227) | 1.194 (3.4709)

3. Secondary Outcome: Mean Change in Transferrin Saturation From Pre-Dialysis to Post-Dialysis
Description: The mean difference between the pre-dialysis and post-dialysis TSAT (transferrin) was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study drug and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
percent
  mean pre-dialysis TSAT (transferrin) | 24.7 (6.67) | 23.2 (8.35)
  mean post-dialysis TSAT (transferrin) | 62.3 (13.32) | 23.3 (7.80)
  pre- to post-dialysis change in TSAT | 37.5 (11.46) | 0.1 (6.87)

4. Secondary Outcome: Mean Change in Unsaturated Iron-Binding Capacity (UIBC) From Pre-Dialysis to Post-Dialysis
Description: The mean difference between the pre-dialysis and post-dialysis unsaturated iron binding capacity (UIBC) was calculated, using all post-baseline values obtained during Stage 2. Subjects could participate in Stage 2 for up to 48 weeks, provided that they did not complete Stage 2 early due to a protocol-mandated change in anemia management or withdraw from the study entirely for other reasons.
Time Frame: Up to 48 weeks from date of randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
micromole per liter
  mean pre-dialysis UIBC | 30.54 (5.645) | 32.19 (6.847)
  mean post-dialysis UIBC | 17.15 (6.030) | 34.75 (7.437)
  pre- to post-dialysis change in UIBC | -13.31 (5.024) | 2.57 (3.345)

5. Secondary Outcome: Red Blood Cell or Whole Blood Transfusion: Number of Patients Who Received a Transfusion
Description: The number of patients requiring red blood cell or whole blood transfusion while in the randomized treatment stage (Stage 2). Patients remained in Stage 2 until they met protocol-defined criteria for Stage 2 completion or until they had participated in Stage 2 for 48 weeks (whichever came sooner). If a patient was transfused, they were withdrawn from Stage 2.
Time Frame: Up to 48 weeks from date of randomization
Population: intent-to-treat: all randomized subjects
Measure: Number; unit: participants
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 147 | 147
participants | 6 | 12

6. Secondary Outcome: Red Blood Cell or Whole Blood Transfusion: Number of Units Transfused
Description: The total number of units of red blood cells or whole blood that were received by patients while in the randomized treatment stage (Stage 2). This number is the total number of units received across all randomized patients in each treatment group (it is not the average number of units received per patient). Patients remained in Stage 2 until they met protocol-defined criteria for Stage 2 completion or until they had participated in Stage 2 for 48 weeks (whichever came sooner). If a patient was transfused, they were withdrawn from Stage 2.
Time Frame: Up to 48 weeks from date of randomization
Population: intent-to-treat: all randomized subjects
Measure: Number; unit: units of red blood cells or whole blood
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 147 | 147
units of red blood cells or whole blood | 15 | 29

7. Secondary Outcome: Percentage of Change From Baseline to End-of-Treatment for: Reticulocyte Hemoglobin Content (CHr), Ferritin, and the Pre-Dialysis Serum Iron Panel
Description: A comparison of the lab values at the end-of-treatment (EoT) to baseline was performed, and the percentage of change from baseline was calculated for the following lab parameters: reticulocyte hemoglobin content (CHr), Ferritin, pre-dialysis unbound iron-binding capacity (UIBC), pre-dialysis serum iron, pre-dialysis transferrin, pre-dialysis total iron-binding capacity TIBC), and transferrin saturation (TSAT).
Time Frame: up to 48 weeks from date of randomization
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
percentage of change from baseline
  CHr percentage of change from baseline | -1.62 (4.402) | -2.59 (4.490)
  Ferritin percentage of change from baseline | -11.6 (29.51) | -21.7 (68.50)
  UIBC percentage of change from baseline | 3.77 (14.717) | 9.46 (16.537)
  Serum Iron percentage of change from baseline | 2.470 (31.3742) | -7.313 (27.8687)
  Transferrin percentage of change from baseline | 1.318 (9.3574) | 3.988 (10.6940)
  TIBC percentage of change from baseline | 1.87 (9.472) | 3.48 (10.166)
  TSAT percentage of change from baseline | 0.6 (29.69) | -10.5 (25.06)

8. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Unsaturated Iron-Binding Capacity (UIBC), Pre-Dialysis Serum Iron, and Pre-Dialysis Total Iron-Binding Capacity (TIBC)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Unsaturated Iron-Binding Capacity (UIBC), Pre-Dialysis Serum Iron, and Pre-Dialysis Total Iron-Binding Capacity (TIBC) will be quantified.
Time Frame: Up to 48 weeks from date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study medication and had at least one post-dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
micromoles per liter
  Baseline UIBC | 30.17 (5.866) | 30.70 (6.481)
  EoT UIBC | 31.03 (6.501) | 33.24 (7.115)
  UIBC Change from Baseline to EoT | 0.92 (4.359) | 2.56 (4.653)
  Baseline Serum Iron | 11.663 (3.7879) | 11.949 (3.9547)
  EoT Serum Iron | 11.438 (3.5804) | 10.658 (3.3615)
  Serum Iron Change from Baseline to EoT | -0.244 (3.4146) | -1.342 (3.3957)
  Baseline TIBC | 41.83 (6.184) | 42.65 (6.942)
  EoT TIBC | 42.47 (6.866) | 43.90 (6.928)
  TIBC Change from Baseline to EoT | 0.67 (0.093) | 1.22 (4.466)

9. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Reticulocyte Hemoglobin (CHr)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Reticulocyte Hemoglobin (CHr)
Time Frame: Up to 48 weeks from date of randomization
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
picograms
  Baseline CHr | 32.57 (2.239) | 32.54 (1.928)
  EoT CHr | 32.01 (2.140) | 31.69 (2.130)
  CHr Change from Baseline to EoT | -0.56 (0.021) | -0.86 (1.480)

10. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Ferritin
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Ferritin
Time Frame: Up to 48 weeks from date of randomization
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: micrograms per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
micrograms per liter
  Baseline Ferritin | 513.6 (201.37) | 479.8 (201.52)
  EoT Ferritin | 446.5 (225.33) | 359.3 (278.61)
  Ferritin Change from Baseline to EoT | -67.1 (164.39) | -122.7 (269.70)

11. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin
Time Frame: Up to 48 weeks from date of randomization
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
grams per liter
  Baseline Transferrin | 1.885 (0.3049) | 1.921 (0.3224)
  EoT Transferrin | 1.902 (0.3267) | 1.987 (0.3366)
  Transferrin Change from Baseline to EoT | 0.019 (0.1839) | 0.066 (0.2138)

12. Secondary Outcome: Change From Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin Saturation (TSAT)
Description: The Mean Change from Stage 2 Baseline to End-of-Treatment (EoT) in Pre-Dialysis Transferrin Saturation (TSAT)
Time Frame: Up to 48 weeks from date of randomization
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
percentage
  Baseline TSAT | 27.9 (8.25) | 28.2 (8.58)
  EoT TSAT | 27.1 (8.01) | 24.6 (8.42)
  TSAT Change from Baseline to EoT | -0.9 (7.65) | -3.7 (7.33)

13. Secondary Outcome: Variability of Hemoglobin Concentration: Temporal Trend
Description: The mean temporal trend of hemoglobin concentration value changes, as measured weekly from baseline until the end of participation in Stage 2.
Time Frame: up to 48 weeks from date of randomization
Population: modified intent-to-treat: all randomized subjects who received at least one dose of study medication and had at least one post dose hemoglobin measured.
Measure: Mean (Standard Deviation); unit: grams per liter per week
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
grams per liter per week | 0.023 (0.222) | 0.003 (0.350)

14. Secondary Outcome: Variability of Hemoglobin Concentration: Residual Standard Deviation
Description: The mean residual standard deviation of the hemoglobin concentration changes, as measured weekly from baseline until the end of participation in Stage 2.
Time Frame: up to 48 weeks from date of randomization
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
grams per liter | 4.352 (1.501) | 4.407 (2.031)

15. Primary Outcome: Change From Baseline Hemoglobin at End-of-Treatment: Mean Baseline and End-of-Treatment Hemoglobin
Description: Mean change from baseline Hgb (the average of the three most recent Hgb values preceding randomization) assessments during the last one-sixth of the treatment period for patients who prematurely withdraw from study treatment, but will include a minimum of at least the last two Hgb values. Values expressed are mean baseline and end-of-treatment Hgb, along with the mean difference (standard deviation).
Time Frame: Hgb measured weekly; up to 48 weeks from date of randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 2 Placebo (Standard Dialysate)
Number analyzed (Participants) | 142 | 144
grams per liter
  Baseline Hemoglobin | 109.6 (6.09) | 109.3 (6.25)
  End-of-Treatment Hemoglobin | 108.7 (13.81) | 104.9 (13.33)
  Mean Change in Hemoglobin from at End-of- | -0.9 (11.76) | -4.5 (11.71)

ADVERSE EVENTS:
Time Frame: In Stage 2, subjects were randomized to placebo or SFP. They were in Stage 2 for up to 48 weeks. Upon completion of Stage 2, subjects could enter the open-label Stage 3 (all received SFP). The maximum total time on study (Stage 2 + Stage 3) was 72 weeks.
Description: The number of subjects included in the safety population = 288, which is 6 subjects fewer than the number of subjects randomized. This discrepancy is due to the fact that the Safety population includes only those subjects exposed to study drug. Six subjects withdrew from Stage 2 prior to study drug exposure.
Groups:
- Stage 2 Standard Dialysate (Placebo): 0 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Standard dialysate: Patients to receive standard dialysate (no iron) during dialysis 3 or 4 times/week in Stage 2 for up to 48 weeks.
- Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate: 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week in Stage 2 for up to 48 weeks.
- Stage 3 Soluble Ferric Pyrophosphate (SFP): 11 micrograms (µg) of iron / deciliter (dL) of dialysate.
  Soluble Ferric Pyrophosphate (SFP): Upon completion of Stage 2, patients to receive 11 micrograms (µg) of iron/ deciliter (dL) of dialysate during dialysis 3 or 4 times/week in Stage 3 for up to 72 weeks of total study participation (Stage 2 + Stage 3).
Arm/Group | Stage 2 Standard Dialysate (Placebo) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate | Stage 3 Soluble Ferric Pyrophosphate (SFP)
Serious Adverse Events (participants affected / at risk) | 36/145 | 44/143 | 83/214
Other Adverse Events (participants affected / at risk) | 93/145 | 89/143 | 179/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2 Standard Dialysate (Placebo) (N=145) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=143) | Stage 3 Soluble Ferric Pyrophosphate (SFP) (N=214)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 (3) | 0 (0) | 4 (4)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
ADVERSE DRUG REACTION (General disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 2 (3) | 0 (0) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
ARTERIOVENOUS FISTULA SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
ARTERIOVENOUS GRAFT SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1) | 8 (8)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CARDIAC ABLATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 2 (2) | 4 (4)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (3) | 4 (5) | 4 (5)
CARDIAC NEOPLASM UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
CATHETER SITE HAEMORRHAGE (General disorders) | 0 (0) | 0 (0) | 2 (2)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
COAGULOPATHY (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
COLONIC POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CONGENITAL CYSTIC KIDNEY DISEASE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED SEPSIS (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
DIABETIC FOOT (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
DIABETIC FOOT INFECTION (Infections and infestations) | 0 (0) | 3 (4) | 2 (2)
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
EXSANGUINATION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 3 (5) | 3 (3) | 10 (12)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
GANGRENE (Infections and infestations) | 0 (0) | 0 (0) | 5 (6)
GASTRIC ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 7 (9)
HYPERPARATHYROIDISM SECONDARY (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1) | 2 (2)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
JOINT ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (2) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (4)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
NECROTISING FASCIITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEUROGLYCOPENIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 2 (2) | 2 (2) | 6 (6)
OBESITY SURGERY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 1 (1) | 3 (5)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 3 (3) | 2 (2) | 4 (5)
POSTERIOR REVERSIBLE ENCEPHALOPATHY SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (5)
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 7 (7)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL CYST HAEMORRHAGE (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
REVERSAL OF ILEOJEJUNAL BYPASS (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SEPSIS SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
STATUS EPILEPTICUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SUDDEN DEATH (General disorders) | 1 (1) | 1 (1) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
TEMPORAL ARTERITIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
VASCULAR GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 2 Standard Dialysate (Placebo) (N=145) | Stage 2 Soluble Ferric Pyrophosphate (SFP) in Dialysate (N=143) | Stage 3 Soluble Ferric Pyrophosphate (SFP) (N=214)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 2 (4) | 9 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5) | 5 (5) | 7 (11)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (8)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 17 (21)
ANGINA PECTORIS (Cardiac disorders) | 2 (3) | 1 (2) | 11 (13)
ANXIETY (Psychiatric disorders) | 3 (3) | 1 (1) | 7 (8)
ARTERIOVENOUS FISTULA SITE COMPLICATION (Injury, poisoning and procedural complications) | 14 (21) | 15 (19) | 52 (85)
ARTERIOVENOUS FISTULA SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 2 (6) | 6 (7) | 12 (18)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 14 (16)
ASTHENIA (General disorders) | 2 (2) | 4 (5) | 17 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (6) | 17 (20)
BRADYCARDIA (Cardiac disorders) | 4 (6) | 4 (10) | 7 (15)
BRONCHITIS (Infections and infestations) | 2 (2) | 5 (5) | 4 (4)
CELLULITIS (Infections and infestations) | 1 (1) | 1 (1) | 7 (7)
CHILLS (General disorders) | 0 (0) | 2 (2) | 8 (13)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 5 (5) | 18 (19)
CONTUSION (Injury, poisoning and procedural complications) | 6 (6) | 6 (6) | 9 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 10 (13) | 18 (23)
DIARRHOEA (Gastrointestinal disorders) | 12 (14) | 10 (12) | 35 (62)
DIZZINESS (Nervous system disorders) | 8 (11) | 9 (19) | 34 (45)
DYSPEPSIA (Gastrointestinal disorders) | 3 (3) | 5 (5) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (11) | 28 (36)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 8 (10)
FACE OEDEMA (General disorders) | 3 (3) | 2 (3) | 12 (15)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 7 (9)
FATIGUE (General disorders) | 4 (4) | 4 (4) | 14 (15)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 7 (8) | 5 (7) | 19 (45)
HAEMODIALYSIS-INDUCED SYMPTOM (Injury, poisoning and procedural complications) | 9 (19) | 10 (14) | 58 (183)
HEADACHE (Nervous system disorders) | 8 (9) | 13 (23) | 40 (61)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 21 (21)
HYPERTENSION (Vascular disorders) | 5 (5) | 5 (6) | 8 (8)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 4 (5) | 5 (5) | 7 (10)
HYPOTENSION (Vascular disorders) | 4 (5) | 5 (5) | 10 (11)
INSOMNIA (Psychiatric disorders) | 5 (5) | 2 (2) | 7 (7)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (8) | 8 (9) | 4 (6)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 8 (9)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 7 (7)
NASOPHARYNGITIS (Infections and infestations) | 9 (11) | 5 (6) | 11 (12)
NAUSEA (Gastrointestinal disorders) | 15 (19) | 11 (21) | 46 (74)
NON-CARDIAC CHEST PAIN (General disorders) | 4 (4) | 2 (2) | 9 (10)
OEDEMA PERIPHERAL (General disorders) | 3 (4) | 12 (14) | 31 (49)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 7 (11)
PAIN (General disorders) | 1 (1) | 1 (1) | 20 (26)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 (12) | 7 (7) | 24 (28)
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 2 (3) | 4 (7) | 8 (20)
PROCEDURAL HEADACHE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 8 (14)
PROCEDURAL HYPERTENSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 12 (26)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 16 (67) | 19 (143) | 75 (567)
PROCEDURAL NAUSEA (Injury, poisoning and procedural complications) | 2 (4) | 1 (1) | 13 (18)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 (2) | 3 (3) | 17 (20)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 10 (10)
PYREXIA (General disorders) | 5 (5) | 5 (5) | 21 (23)
TACHYCARDIA (Cardiac disorders) | 4 (5) | 1 (14) | 8 (11)
THROMBOSIS IN DEVICE (General disorders) | 0 (0) | 2 (2) | 8 (14)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 3 (3) | 7 (10)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8) | 8 (11) | 12 (16)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 5 (7) | 6 (6)
VASCULAR GRAFT COMPLICATION (Injury, poisoning and procedural complications) | 4 (8) | 2 (3) | 11 (13)
VASCULAR GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 7 (8)
VOMITING (Gastrointestinal disorders) | 12 (16) | 11 (15) | 33 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less